CLINICAL TRIAL: NCT04075552
Title: Improving Healthy Eating of Children With Autism in a School Setting
Brief Title: Healthy Eating ASD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Disruptions due to COVID-19
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jonathan Ivy, Assistant Professor of Psychology, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005814
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Food Selectivity

STUDY DESIGN:
Intervention Model Description: Single subject research methodology
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants are students from a specialized school for children with autism.
  Interventions: Behavioral: Pre Meal Presentation; Behavioral: Pre Meal Presentation + Modeling; Behavioral: Pre Meal Presentation + Token Economy

INTERVENTIONS:
Behavioral: Pre Meal Presentation — Pre-Meal Presentation. In the Pre-Meal Presentation (PMP) condition, school staff delivered the plate of vegetable pieces prior to students regularly scheduled lunchtime (about 5 min). Like baseline, no programmed consequences were provided for student interaction or consumption of the vegetables.
Behavioral: Pre Meal Presentation + Modeling — Similar to the prior condition, each participant will be offered a plate containing target foods for 4 min. Once the plate has been delivered to each participant, a staff person will model eating the food. The model will have an identical plate of food. Within six feet of students oriented towards the model (i.e., the students will be facing the model), the model will pick up one piece of food, say "Yum, this looks good" in a loud and excited tone, eat it, and then deliver a "soft" prompt to the participants to try it (e.g., "You should try this!"). Staff will avoid giving a firm/hard demand (e.g., "Eat the food"). Repeat this for four pieces of food, alternating between the two target foods, with about 10-20 sec between each bite. Repeat the model as necessary based on the room arrangement, such that each students contacts the model within six feet while oriented towards the model.
Behavioral: Pre Meal Presentation + Token Economy — Similar to prior condition, expect each participant can earn tokens for eating food items. Tokens can be exchanged for small prizes (e.g., pencil or sticker) at the end of a session.

SUMMARY:
Most studies which have addressed food selectivity among children with autism spectrum disorders have been conducted in either clinic or home settings. School-based research has been conducted to increase healthy eating, but this research was largely conducted with children without special needs or if children with special needs did participate, they were not identified.

This study will focus on increasing consumption of fruits and vegetables among children with an Autism Spectrum Disorder in a school setting.

DETAILED DESCRIPTION:
Food Preference Inventory: A survey of food preference and eating habits, developed by the experimenter, will be provided to the parents/guardians of prospective participants. The Food Preference Inventory is anticipated to take between 10 and 20 mins to complete. The parent/guardian of the prospective participant is asked to return toe inventory to the school if 1) the parent/guardian gives permission for his/her child to participate and 2) if the child does not have a food allergy.

General Procedures: Each day of the study (1-5 days per week), school staff will offer participants a small portion of a fruit or vegetable (about 1/8 cup) to eat during lunch time. The participant will have about 5 min to consume the item before it is recollected by school staff.

Baseline: The fruit or vegetable is presented with the participants lunch. Eating the item produces no programmed consequences.

Single Item Presentation: The fruit or vegetable is presented before the participants lunch (about 5 min). Eating the item produces no programmed consequences.

Single Item Presentation + Modeling: The fruit or vegetable is presented before the participants lunch (about 5 min). School staff will model eating the food item.

Single Item Presentation + Token Economy: The fruit or vegetable is presented before the participants lunch (about 5 min). Eating the item will produce a token (e.g., a sticker or hole punch). Once the student collects a few tokens (e.g., 3-5), he/she can exchange the tokens for a small price (e.g., pencil or crayon).

Data Collection: Data will be collected by school staff. Staff will record whether each participant consume the fruit or vegetable item.

Safety Procedures: School staff will monitor lunch - as they typically do.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be students in a private school with a diagnosis of an autism spectrum disorder and between 6-14 years of age.

Exclusion Criteria:

* Parents who report their children have food allergies of any kind will be excluded.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Increased consumption of healthy foods | Through study completion, 1 year.
  Direct measure of the number of healthy foods items eaten

CONTACTS AND LOCATIONS:
Locations (1):
- Hogan Learning Academy, Fleetwood, Pennsylvania, United States